CLINICAL TRIAL: NCT06364696
Title: An Open-label Phase 1 Study of ASP4396 in Participants With Locally Advanced (Unresectable) or Metastatic Solid Tumor Malignancies With KRAS G12D Mutation
Brief Title: A Study to Find a Suitable Dose of ASP4396 in Adults With Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4396-CL-0101
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor
Keywords: Locally Advanced Solid Tumors; Metastatic Solid Tumors; ASP4396; KRAS G12D; Non-small Cell Lung Cancer; Colorectal Cancer; Pancreatic Ductal Adenocarcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ASP4396 Dose Escalation (Experimental): Participants will receive ASP4396 in a 21-day cycle.
  Interventions: Drug: ASP4396
- ASP4396 Dose Expansion (Experimental): Participants will receive ASP4396 in a 21-day cycle.
  Interventions: Drug: ASP4396

INTERVENTIONS:
Drug: ASP4396 — Intravenous (IV) infusion

SUMMARY:
Genes contain genetic code which tell the body which proteins to make. Some types of cancer are caused by changes, or mutations, in a gene called KRAS. Researchers are looking for ways to stop the actions of abnormal proteins made from the mutated KRAS gene. The so-called G12D mutation in the KRAS gene is common in people with some solid tumors.

ASP4396 is being developed as a potential new treatment for solid tumors in people who have the G12D mutation in their KRAS gene. ASP4396 is not currently available as a treatment for the public. In this study, researchers will learn how ASP4396 is processed by and acts upon the body. This information will help find a suitable dose and to check for potential medical problems from ASP4396.

In this study, ASP4396 is being given to humans for the first time.

People in this study will be adults with locally advanced (unresectable), or metastatic solid tumors with the G12D mutation in their KRAS gene. Locally advanced means the cancer has spread to nearby tissue. Unresectable means the cancer cannot be removed by surgery. Metastatic means the cancer has spread to other parts of the body. They may have been previously treated with standard therapies or refused to receive those treatments.

The main aims of the study are to check the safety of ASP4396, how well people cope with medical problems during the study (how well it is tolerated), and to find a suitable dose of ASP4396.

This is an open-label study. This means that people in this study and clinic staff will know that they will receive ASP4396.

This study will be in 2 parts.

Part 1 is called Dose Escalation. Different small groups of people will receive lower to higher doses of ASP4396. For each dose, all medical problems will be recorded. The first group will receive the lowest dose of ASP4396. A medical expert panel will check the results and decide if the next group can receive a higher dose of ASP4396. The panel will do this until all groups have taken ASP4396 or until suitable doses have been selected for Part 2.

Part 2 is called Dose Expansion. Other different small groups of people will receive ASP4396 with the most suitable doses worked out from Part 1. This will help find a more accurate dose of ASP4396 to use in future studies.

In both parts of the study, ASP4396 will be given through a vein. This is called an infusion. Each treatment cycle is 21 days long. People will continue treatment until: they have medical problems from the treatment they can't cope with (can't tolerate); their cancer gets worse; they start other cancer treatment; or they ask to stop treatment.

People will visit the clinic on certain days during their treatment, with extra visits during the first 2 cycles of treatment. The study doctors will check for any medical problems from ASP4396. Also, people in the study will have a health check including blood tests. On some visits they will also have scans to check for any changes in their cancer. Tumor samples will be taken at certain visits during treatment with the option of a tumor sample being taken after treatment has finished.

People will visit the clinic about 7 days after they stop treatment. They will be asked about any medical problems and will have a health check including blood tests.

After this, people will visit the clinic for a health check several times. The number of visits and checks done at each visit will depend on the health of each person and whether they completed their treatment or not.

After treatment has finished, people in the study will be followed up for up to 45 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant has locally advanced (unresectable) or metastatic solid tumor malignancy with documented KRAS G12D mutation and has received prior standard therapy.
* Participant has at least 1 measurable lesion per RECIST v1.1.
* Participant has an ECOG performance status of 0 or 1.
* Participant has adequate organ function.

Exclusion Criteria:

* Participant has symptomatic or untreated central nervous system (CNS) metastases. Participants with asymptomatic and treated and stable CNS metastases are eligible.
* Participant has leptomeningeal disease as a manifestation of the current malignancy.
* Participant has another prior malignancy active (i.e., requiring treatment or intervention) within the previous 2 years different from the primary malignancy for this study, except for local malignancies that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast, which are allowed.
* Participant with active hepatitis B or hepatitis C virus (HCV).
* Participant has a known history of human immunodeficiency virus (HIV) infection with acquired immunodeficiency syndrome (AIDS)-related complications.
* Participant has an active infection requiring intravenous antibiotics within 14 days prior to study intervention.
* Participant is expected to require another form of anticancer therapy while on study intervention.
* Participant has any condition that makes the participant unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) for ASP4369 | Up to 21 days
  A DLT is defined as any event meeting the DLT criteria occurring within 21 days of first dose on Cycle 1 at least possibly related to study intervention.
Number of Participants with Adverse Events (AEs) | Up to 12 months
  An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants with Serious Adverse Events (SAEs) | Up to 12 months
  An SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and other medically important events.
Number of Participants with laboratory value abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant laboratory values.
Number of Participants with electrocardiogram (ECG) abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant ECG values.
Number of Participants with vital sign abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant vital sign values.
Number of Participants with physical exam abnormalities and/or AEs | Up to 12 months
  Number of participants with potentially clinically significant physical exam values or symptoms.
Number of Participants with Eastern Cooperative Oncology Group (ECOG) performance status score | Up to 12 months
  The ECOG scale will be used to assess performance status. Grades range from 0 (fully active) to 5 (dead). Negative change scores indicate an improvement. Positive scores indicate a decline in performance.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 12 months
  ORR is defined as the proportion of participants whose best overall response with confirmation status is rated as (confirmed or unconfirmed) complete response (CR) or (confirmed or unconfirmed) partial response (PR) based on RECIST v1.1.
Duration of Response (DOR) per RECIST v 1.1 | Up to 12 months
  DOR is measured from the day the criteria are first met for time point overall response rated as CR or PR (whichever is first recorded) until the first date of documented radiological disease progression per RECIST v1.1 or death in the absence of progression.
Disease Control Rate (DCR) per RECIST v 1.1 | Up to 12 months
  DCR is defined as the proportion of participants whose best overall response with confirmation status is rated as (confirmed or unconfirmed) CR, (confirmed or unconfirmed) PR or stable disease (SD) (including non-CR/non-progressive disease [PD] for participants with no measurable disease at baseline) based on RECIST v1.1.
Progression Free Survival (PFS) per RECIST v1.1 | Up to 12 months
  PFS is defined as the time from the start of study intervention until the date of documented radiological disease progression per RECIST v1.1 or until death for any cause, whichever comes first.
Overall Survival (OS) | Up to 12 months
  OS is defined as the time from the start of study intervention until death due to any cause.
Pharmacokinetics (PK) of ASP4396 in plasma: area under the concentration-time curve from the time of dosing to 24 hours after dosing (AUC24h) | Up to 12 months
  AUC24h will be recorded from the PK plasma samples collected.
PK of ASP4396 metabolite in plasma: AUC24h | Up to 12 months
  AUC24h will be recorded from the PK plasma samples collected.
PK of ASP4396 in plasma: AUC168h | Up to 12 months
  AUC168h will be recorded from the PK plasma samples collected.
PK of ASP4396 metabolite in plasma: AUC168h | Up to 12 months
  AUC168h will be recorded from the PK plasma samples collected.
PK of ASP4396 in plasma: Maximum Concentration (Cmax) | Up to 12 months
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP4396 metabolite in plasma: Cmax | Up to 12 months
  Cmax will be recorded from the PK plasma samples collected.
PK of ASP4396 in plasma: concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to 12 months
  Ctrough will be recorded from the PK plasma samples collected.
PK of ASP4396 metabolite in plasma: Ctrough | Up to 12 months
  Ctrough will be recorded from the PK plasma samples collected.
PK of ASP4396 in plasma: Time of maximum concentration (tmax) | Up to 12 months
  tmax will be recorded from the PK plasma samples collected.
PK of ASP4396 metabolite in plasma: tmax | Up to 12 months
  tmax will be recorded from the PK plasma samples collected.
Change from baseline of Kirsten rat sarcoma viral oncogene homolog (KRAS) G12D amino acid substitution (G12D) tumor samples | Baseline and up to 12 months
  Changes in KRAS G12D in tumor samples will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma Inc
Locations (7):
- United States (7):
  - University of Kansas Cancer Center, Westwood, Kansas
  - START Midwest, Grand Rapids, Michigan
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester, Rochester, New York
  - NEXT Oncology Dallas, Irving, Texas
  - START Mountain Region, West Valley City, Utah
  - NEXT Oncology Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/